CLINICAL TRIAL: NCT01051232
Title: A Double Blind, Placebo-Controlled, Randomized, Dose Escalation Study To Investigate Safety, Tolerability, And Pharmacokinetics Of PF-00868554 (Filibuvir) Following Single Oral Administrations Of PF-00868554 (Filibuvir) Under Fasting Conditions In Japanese Healthy Adult Volunteers
Brief Title: A Study To Investigate Safety And Pharmacokinetics Of A Single Dose Of PF-00868554 (Filibuvir) In Japanese Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: A8121035
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: filibuvir; pharmacokinetics; Japanese; Asian
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Placebo Comparator): PF-00868554 (filibuvir) 100 mg or placebo
  Interventions: Drug: Active; Drug: Placebo
- Cohort 2 (Placebo Comparator): PF-00868554 (filibuvir) 300 mg or placebo
  Interventions: Drug: Active; Drug: Placebo
- Cohort 3 (Placebo Comparator): PF-00868554 (filibuvir) 500 mg or placebo
  Interventions: Drug: Active; Drug: Placebo

INTERVENTIONS:
Drug: Active — Six subjects will receive PF-00868554 (filibuvir) 100 mg under fasting condition.
  Arms: Cohort 1
Drug: Placebo — Two subjects will receive the placebo under fasting condition.
  Arms: Cohort 1
Drug: Active — Six subjects will receive PF-00868554 (filibuvir) 300 mg under fasting condition.
  Arms: Cohort 2
Drug: Placebo — Two subjects will receive the placebo under fasting condition.
  Arms: Cohort 2
Drug: Active — Six subjects will receive PF-00868554 (filibuvir) 500 mg under fasting condition.
  Arms: Cohort 3
Drug: Placebo — Two subjects will receive the placebo under fasting condition.
  Arms: Cohort 3

SUMMARY:
A single dose of PF-00868554 (filibuvir) will be safety and tolerable in Japanese healthy volunteers. The pharmacokinetics in Japanese will be consistent to that available in Western population.

DETAILED DESCRIPTION:
Investigation of safety, tolerability and pharmacokinetics of single oral administration of PF-00868554 (filibuvir) in healthy adult Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 20 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg.

Exclusion Criteria:

* A positive result for Hepatitis B surface antigen (HbsAg) or anti-hepatitis C virus serology, and HIV antigen/antibody.
* Male subjects with a history of subfertility/infertility and other conditions that in the opinion of the investigator may affect fertility.
* Pregnant or nursing females; females of childbearing potential.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety; ECGs/vital signs | Screening to Follow-up (Day 5)
Safety; laboratory tests | Screening to Follow-up (Day 5)
Safety; physical examination/adverse event monitoring | Screening to Follow-up (Day 5)

SECONDARY OUTCOMES:
Pharmacokinetics; Plasma PF-00868554 (filibuvir) concentrations | Day 1 to Day 3
Pharmacokinetics; Urine PF-00868554 (filibuvir) concentrations | Day 1 to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121035&StudyName=A%20Study%20To%20Investigate%20Safety%20And%20Pharmacokinetics%20Of%20A%20Single%20Dose%20Of%20PF-00868554%20%28Filibuvir%29%20In%20Japanese%20Healthy%20Adult%20Volunteers